CLINICAL TRIAL: NCT01373242
Title: Peanut Sublingual Immunotherapy and Induction of Clinical Tolerance in Peanut Allergic Children (SLIT Tolerance TLC) {Sublingual Immunotherapy for Peanut Allergy}
Brief Title: Sublingual Immunotherapy for Peanut Allergy and Induction of Tolerance
Acronym: SLIT-TLC
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-2308; 5R01AT004435-09 (NIH)
Record Dates: First submitted 2011-06-12; First posted 2011-06-14 (Estimated); Results first posted 2019-06-12 (Actual); Last update posted 2019-06-12 (Actual); Status verified 2018-10

CONDITIONS: Peanut Hypersensitivity; Food Hypersensitivity; Food Allergy; Peanut Allergy
MeSH Terms: conditions — Peanut Hypersensitivity; Food Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Peanut ( liquid peanut extract) SLIT (Experimental): All subjects will receive peanut SLIT upon enrollment for at least the first 48 months. After the desensitization DBPCFC after at least 48 months of treatment, subjects will be randomized off treatment from 1 to 17 weeks. Subjects will then undergo another DBPCFC.
  Interventions: Drug: Liquid peanut extract (Peanut SLIT)

INTERVENTIONS:
Drug: Liquid peanut extract (Peanut SLIT) — Liquid peanut extract will be administered under the tongue
  Other Names: Peanut SLIT - active arm

SUMMARY:
The goal of this study will be to increase the reaction threshold (desensitization) of peanut allergic children using peanut sublingual immunotherapy and to determine if the nonreactive state of the immune system persists after treatment has been discontinued (tolerance).

DETAILED DESCRIPTION:
Allergy to peanuts and tree nuts affects approximately 1.4% of the population. Allergic reactions to peanut can be severe and life threatening and account for the vast majority of fatalities due to food-induced anaphylaxis. At present, there are no viable treatment options for patients with peanut allergy. The current standard of care is strict dietary elimination and emergency preparedness with an anaphylaxis kit in the event of an accidental reaction.

Our group and others have shown that oral immunotherapy can provide protection from anaphylaxis to a variety of food proteins. In addition, our ongoing research has demonstrated that sublingual immunotherapy to peanut provides a safe, alternative mode of immunotherapy to reduce allergic reaction rates (desensitization) during oral food challenge (OFC) to peanut. The goal of this study will be to desensitize peanut allergic children using peanut sublingual immunotherapy and to determine if the nonreactive state of the immune system persists after treatment has been discontinued (tolerance). Children ages 1-11 years will be enrolled following an entry double blind, placebo controlled food challenge (DBPCFC).

After at least 48 months of peanut SLIT study drug, subjects will undergo a second DBPCFC to 5000 mg of peanut protein to assess desensitization.

* Subjects who are not desensitized are those who are not able to consume more than the MCRT without symptoms, which has been defined as 300 mg of peanut protein. Subjects who consume less than 300 mg of peanut protein without symptoms will stop peanut SLIT and conclude the study. These subjects will not undergo any additional study procedures including the remaining protocol DBPCFCs and will be recommended to resume a strict peanut avoidance diet.
* Subjects who are able to consume more than 300 mg of peanut protein will be randomized to an interval between 1 and 17 weeks during which all peanut including peanut SLIT study drug will be discontinued. This period of avoidance will be followed by a third DBPCFC to 5000 mg of peanut protein to evaluate for the loss of the desensitization effect. After this final DBPCFC, the study will be completed for these subjects. At the primary investigators clinical discretion, they will be recommended to transition to a daily peanut food equivalent to maintain the desensitized effect.

Outcome variables of interest include response to double blind, placebo controlled food challenges, skin prick testing, peanut specific serum immunoglobin E (IgE), immunoglobin G (IgG), and immunoglobin G4 (IgG4) and salivary immunoglobin A (IgA), T and B cell responses, basophil hyporesponsiveness, quality of life, and adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Between ages 1 year to 12 years exclusive
* Peanut specific IgE > 0.35kU/L or a convincing clinical history of an allergic reaction to peanut within 1 hour of ingestion
* Positive entry DBPCFC to 1 gram of peanut protein

Exclusion Criteria:

* History of severe anaphylaxis to peanut, defined as hypoxia, hypotension, or neurologic compromise (cyanosis or oxygen saturations < 92% at any stage, hypotension, confusion, collapse, loss of consciousness, or incontinence)
* Participation in any interventional study for the treatment of food allergy in the past 6 months
* Known oat, wheat, or glycerin allergy
* Eosinophilic or other inflammatory (e.g. celiac) gastrointestinal disease
* Severe asthma (2007 National Heart Lung and Blood Institute (NHLBI) guidelines Criteria Steps 5 or 6 - Appendix 2)
* Inability to discontinue antihistamines for skin testing and DBPCFCs
* Use of omalizumab or other non-traditional forms of allergen immunotherapy (e.g., oral or sublingual) or immunomodulator therapy (not including corticosteroids) or biologic therapy within the past year
* Use of beta-blockers (oral), angiotensin-converting enzyme (ACE) inhibitors, angiotensin-receptor blockers (ARB) or calcium channel blockers
* Significant medical condition (e.g., liver, kidney, gastrointestinal, cardiovascular, hematologic, or pulmonary disease) which would make the subject unsuitable for induction of food reactions

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 54 (Actual)
Dates: Start 2011-06 (Actual); Primary Completion 2018-04-16 (Actual); Study Completion 2018-04-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wesley Burks, MD, Principal Investigator — University of North Carolina
Locations (1):
- University of North Carolina, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Peanut allergic children ages 1-11 years
Groups:
- Peanut (Liquid Peanut Extract) SLIT: All subjects will receive peanut SLIT upon enrollment for at least 48 months and then undergo a desensitization DBPCFC. Subjects will then be randomized to be off treatment for a period between 1 to 17 weeks. Subjects will then undergo a final DBPCFC.
  Liquid peanut extract (Peanut SLIT): Liquid peanut extract will be administered under the tongue
Period: Overall Study
Arm/Group | Peanut (Liquid Peanut Extract) SLIT
Started | 54
Completed | 38
Not Completed | 16

BASELINE CHARACTERISTICS:
Arm/Group | Peanut ( Liquid Peanut Extract) SLIT
Number analyzed (Participants) | 54
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 54
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] — Inclusion criteria: age 1 year up to but not including 12 years.
  years | 7.05 [2.3 to 11.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 34
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 49
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 54
Peanut-specific IgE (kU/L) [Median (Full Range); unit: kU/L] | 85.6 [0.3 to 1804]
Peanut skin prick test wheal size (mm) [Median (Full Range); unit: mm] | 16 [2 to 36.5]

OUTCOME MEASURES:

1. Primary Outcome: Population Sensitization Threshold in mg Peanut Protein Predicted to Provoke Reactions in 5% of the Peanut-allergic Population
Description: An estimate of the dose as assessed by the 48th month DBPCFC reported in mg peanut protein, also called population sensitization threshold, predicted to provoke reactions in 5% of the peanut-allergic population. This will also give population level no observed adverse event level (NOAEL) and lowest observed adverse event level (LOAEL) that would define interval of consecutive administered dose levels within which the population sensitization threshold lies. NOAEL is the highest dose observed not to produce any adverse effect and LOAEL is the lowest dose that is observed to produce an adverse effect.
Time Frame: 48 - 52 months
Measure: Number; unit: mg
Arm/Group | Peanut (Liquid Peanut Extract) SLIT
Number analyzed (Participants) | 54
mg
  NOAEL threshold | 160
  LOAEL threshold | 300

2. Primary Outcome: Population Sensitization Threshold in mg Peanut Protein Predicted to Provoke Reactions in 10% of the Peanut-allergic Population
Description: An estimate of the dose as assessed by the 48th month DBPCFC reported in mg peanut protein, also called population sensitization threshold, predicted to provoke reactions in 10% of the peanut-allergic population. This will also give population level no observed adverse event level (NOAEL) and lowest observed adverse event level (LOAEL) that would define interval of consecutive administered dose levels within which the population sensitization threshold lies. NOAEL is the highest dose observed not to produce any adverse effect and LOAEL is the lowest dose that is observed to produce an adverse effect.
Time Frame: 48-52 months
Measure: Number; unit: mg
Arm/Group | Peanut (Liquid Peanut Extract) SLIT
Number analyzed (Participants) | 54
mg
  NOAEL threshold | 800
  LOAEL threshold | 750

3. Primary Outcome: Population Estimate of Time for a Subject's True Sensitivity Threshold to Reduce by Half.
Description: A population estimate of time to loss of desensitization will be calculated for a subject's true sensitivity threshold (LOAEL) to reduce by half, also called half-life of sensitivity threshold. This is calculated based on the Kaplan-Meier estimator of the survival function using study participant data.
Time Frame: 52 months
Measure: Number; unit: weeks
Arm/Group | Peanut (Liquid Peanut Extract) SLIT
Number analyzed (Participants) | 54
weeks | 17

4. Primary Outcome: Population Estimate of a Subject's True Sensitivity Threshold to Maintain at the Same Dose Level During DBPCFC
Description: A population estimate of time to loss of desensitization will be calculated for a subject's true sensitivity threshold (LOAEL) to maintain at the same dose level during the double-blind, placebo-controlled food challenge. Food challenge dose levels are as follows: 100 mg, 200 mg, 500 mg, 800 mg, 1300 mg, 2100 mg. This is calculated based on the Kaplan-Meier estimator of the survival function using study participant data.
Time Frame: 52 months
Measure: Number; unit: weeks
Arm/Group | Peanut (Liquid Peanut Extract) SLIT
Number analyzed (Participants) | 54
weeks | 13

5. Primary Outcome: Population Estimate of a Subject's True Sensitivity Threshold to Decrease by One Dose Level of During the DBPCFC
Description: A population estimate of time to loss of desensitization will be calculated for a subject's true sensitivity threshold (LOAEL) to decrease by one dose level during the double-blind, placebo-controlled food challenge. Food challenge dose levels are as follows: 100 mg, 200 mg, 500 mg, 800 mg, 1300 mg, 2100 mg. This is calculated based on the Kaplan-Meier estimator of the survival function using study participant data.
Time Frame: 52 months
Measure: Number; unit: weeks
Arm/Group | Peanut (Liquid Peanut Extract) SLIT
Number analyzed (Participants) | 54
weeks | 14

6. Secondary Outcome: Number of Participants With Adverse Events and Serious Adverse Events During the Study.
Description: Number of participants with adverse events (AEs) and serious adverse events (SAEs) during the SLIT treatment portion of the study.
Time Frame: 48 months
Measure: Count of Participants; unit: Participants
Arm/Group | Peanut (Liquid Peanut Extract) SLIT
Number analyzed (Participants) | 54
Participants
  Adverse events | 53
  Serious adverse events | 0

7. Secondary Outcome: Number of Participants With Gastrointestinal and Possible Gastrointestinal Eosinophilic Adverse Events.
Description: With published concerns for the development of eosinophilic gastrointestinal disease after food immunotherapy, will report the number of participants with gastrointestinal and possible gastrointestinal eosinophilic adverse events during SLIT therapy
Time Frame: 48 months
Measure: Count of Participants; unit: Participants
Arm/Group | Peanut (Liquid Peanut Extract) SLIT
Number analyzed (Participants) | 54
Participants
  Gastrointestinal adverse events | 16
  Possible eosinophilic gastrointestinal AEs | 2

8. Secondary Outcome: Change in Peanut Skin Test Wheal Over Time Among Subjects Who Were Induced With Clinical Desensitization Versus Those Who Failed
Description: Comparative estimates of changes in immune parameters (wheal size in mm during peanut skin prick test) from baseline through end of treatment among subjects who were induced with clinical desensitization (ingesting 5000mg on DBPCFC without symptoms) versus those who failed (developing clinical symptoms after ingesting 5000mg on DBPCFC).
Time Frame: 48 months
Measure: Median (Full Range); unit: mm
Groups:
- Desensitized After Peanut SLIT: All subjects will receive peanut SLIT upon enrollment for at least 48 months and then undergo a desensitization DBPCFC. 'Desensitized' defined as completing the 5000mg desensitization DBPCFC without dose limiting symptoms.
- Non-desensitized After Peanut SLIT: All subjects will receive peanut SLIT upon enrollment for at least 48 months and then undergo a desensitization DBPCFC. 'Non-desensitized' defined as experiencing dose limiting symptoms during the 5000mg desensitization DBPCFC.
Arm/Group | Desensitized After Peanut SLIT | Non-desensitized After Peanut SLIT
Number analyzed (Participants) | 17 | 37
mm
  Baseline wheal size | 14.5 [2 to 27] | 16.25 [5.5 to 36.5]
  48 month wheal size | 7.25 [1 to 14] | 9.25 [2 to 25.5]

9. Secondary Outcome: Change in Peanut IgE Over Time Among Subjects Who Were Induced With Clinical Desensitization Versus Those Who Failed
Description: Comparative estimates of changes in immune parameters (serum levels of peanut specific IgE in kU/L) from baseline through end of treatment among subjects who were induced with clinical desensitization (ingesting 5000mg on DBPCFC without symptoms) versus those who failed (developing clinical symptoms after ingesting 5000mg on DBPCFC).
Time Frame: 48 months
Measure: Median (Full Range); unit: kU/L
Arm/Group | Desensitized After Peanut SLIT | Non-desensitized After Peanut SLIT
Number analyzed (Participants) | 17 | 37
kU/L
  Baseline peanut IgE | 107 [0.3 to 1139.4] | 84.7 [10.9 to 1804]
  48 month peanut IgE | 12.1 [0.05 to 484] | 11.2 [1.4 to 970]

10. Secondary Outcome: Change in Peanut IgG4 Over Time Among Subjects Who Were Induced With Clinical Desensitization Versus Those Who Failed
Description: Comparative estimates of changes in immune parameters (serum levels of peanut-specific IgG4 in mg/L) from baseline through end of treatment among subjects who were induced with clinical desensitization (ingesting 5000mg on DBPCFC without symptoms) versus those who failed (developing clinical symptoms after ingesting 5000mg on DBPCFC).
Time Frame: 48 months
Measure: Median (Full Range); unit: mg/L
Arm/Group | Desensitized After Peanut SLIT | Non-desensitized After Peanut SLIT
Number analyzed (Participants) | 17 | 37
mg/L
  Baseline peanut IgG4 | 0.47 [0.02 to 6.38] | 0.37 [0.02 to 19.65]
  48 month peanut IgG4 | 9.69 [0.04 to 80] | 4.39 [0.05 to 57.4]

ADVERSE EVENTS:
Time Frame: Adverse event data collected over 48 month peanut SLIT treatment period.
Arm/Group | Peanut (Liquid Peanut Extract) SLIT
All-Cause Mortality (participants affected / at risk) | 0/54
Serious Adverse Events (participants affected / at risk) | 0/54
Other Adverse Events (participants affected / at risk) | 53/54
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Peanut (Liquid Peanut Extract) SLIT (N=54)
Vomiting (Gastrointestinal disorders) | 8
Diarrhea (Gastrointestinal disorders) | 3
Rash (Skin and subcutaneous tissue disorders) | 4
Runny nose (Respiratory, thoracic and mediastinal disorders) | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2
Oropharyngeal itch (Skin and subcutaneous tissue disorders) | 36
Sneezing (Respiratory, thoracic and mediastinal disorders) | 3
Coughing (Respiratory, thoracic and mediastinal disorders) | 3
Itchy nose (Skin and subcutaneous tissue disorders) | 1
Skin itch (Skin and subcutaneous tissue disorders) | 14
Lip swelling (Skin and subcutaneous tissue disorders) | 15
Eye swelling (Skin and subcutaneous tissue disorders) | 2
Eye itch (Skin and subcutaneous tissue disorders) | 2
Eye tearing (Skin and subcutaneous tissue disorders) | 2
Hives (Skin and subcutaneous tissue disorders) | 10
Belly pain (Gastrointestinal disorders) | 16
Nasal congestion (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-03-02): https://cdn.clinicaltrials.gov/large-docs/42/NCT01373242/Prot_000.pdf
  • Statistical Analysis Plan (2016-02-13): https://cdn.clinicaltrials.gov/large-docs/42/NCT01373242/SAP_001.pdf